CLINICAL TRIAL: NCT00435500
Title: Fluoride Varnish in the Prevention of Dental Caries in Aboriginal and Non-aboriginal Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOP-64215
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Dental Caries
Keywords: Dental caries, topical fluorides
MeSH Terms: conditions — Dental Caries

INTERVENTIONS:
Drug: Fluoride varnish

SUMMARY:
The purpose of this study is to determine whether semi-annual fluoride varnish applications combined with caregiver counseling are effective in preventing and reducing a severe form of dental decay, known as early childhood caries, in native and non-native children aged 6 months to 5 years.

DETAILED DESCRIPTION:
Early childhood caries (ECC) is by far the most common chronic disease among Canadian Aboriginal children, affecting nearly 90% of First Nations preschoolers in Ontario. It is the number one cause of oral health disparities between native and non-native children. ECC negatively impacts on the quality of life of children suffering from the disease and the caregivers and family members who care for them. To address the problem of ECC, a range of health promotion campaigns, including parent education aimed at balancing the knowledge and values of First Nations communities with the recommendations of the scientific community, have been implemented but these initiatives have had limited success in reducing the impact of ECC and its treatment.

While oral health promotion campaigns have raised awareness of the severity of ECC among these communities, the literature shows that for this age cohort, increasing host resistance through professionally applied topical fluoride (PATF) applications at regular intervals may achieve better results. Of all the PATF methods, slow-release fluoride varnish may be the most practical alternative to the use of gels, foams and rinses, as it decreases the risk of fluoride ingestion and is associated with greater patient acceptability. Fluoride varnish has shown promise as a caries reduction agent but more evidence for the effectiveness of this intervention is needed, particularly for high-caries-risk populations like those in Aboriginal communities.

The aim of this study is to determine the effectiveness of fluoride varnish (Duraflor, 5% NaF, Pharmascience) combined with caregiver counseling in preventing and reducing ECC in Aboriginal communities, in a 2-year randomized controlled trial. Methods: The trial enrolled 1226 children aged 6 months to 5 years from the Sioux Lookout Zone (SLZ) First Nations reserves and 149 from Thunder Bay (NW Ontario). Twenty First Nations communities were randomized to 2 study groups; families in both groups received oral health counseling and restorative dental care provided by the SLZ Dental Program - one group received no fluoride varnish (FV0) and the other received FV 2-3×/yr. The same subjects were examined for the dmft/s indices by trained and calibrated dental hygienists in 2003, 2004 and 2005. A caregiver questionnaire assessed the impact of ECC on the quality of life of the child and the family. The SLZ Hospital provided data on children's dental general anesthetic (GA) procedures. Comparative cross-sectional oral health data for 416 (2003), 687 (2004) and 544 (2005) 3-5 yr-olds attending Junior Kindergarten in Thunder Bay, not receiving fluoride treatments, were collected by the Thunder Bay District Health Unit's dental hygienists and recorders. Results will assist decision makers in developing programs for addressing the problem of ECC in high-caries-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least one primary tooth present.
* Age 6 months to <6 years. Children under 6 months of age may be enrolled in the study if at least one primary tooth has erupted.
* Residing in one of the First Nations Communities in the Sioux Lookout Zone or in the Thunder Bay District Area, both located in Northwestern Ontario, Canada.
* Parental consent must be provided. If the parent is not the primary caregiver, a legal guardian or a family member who is the primary care provider must sign the consent form.

Exclusion Criteria:

* Children with ulcerative gingivitis and stomatitis. (These children will be referred for treatment.)
* Children with allergy to colophony (colophonium). Colophonium is found in some cosmetics, creams, sunscreens, pine-oil cleaners, chewing gum, and postage stamp glue. Parents will be asked if the child suffers from this particular allergy.
* No teeth present or stainless steel crowns only.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1320
Dates: Start 2003-06; Study Completion 2006-01

PRIMARY OUTCOMES:
Reduction in the 2-year caries increment (dmfs/DMFS index); final follow-up at 24 months.

SECONDARY OUTCOMES:
(1) Need for dental treatment under general anaesthesia at 24 months; (2) score on an oral-health-related quality of life scale at 24 months; (3) the annualized cost of fluoride varnish treatment per child

CONTACTS AND LOCATIONS:
Overall Officials: Herenia P. Lawrence, DDS, PhD, Principal Investigator — University of Toronto, Faculty of Dentistry, Toronto, Ontario, Canada
Locations (1):
- Sioux Lookout Zone Dental Program, Sioux Lookout, Ontario, Canada

REFERENCES:
- [Derived] Lawrence HP, Binguis D, Douglas J, McKeown L, Switzer B, Figueiredo R, Laporte A. A 2-year community-randomized controlled trial of fluoride varnish to prevent early childhood caries in Aboriginal children. Community Dent Oral Epidemiol. 2008 Dec;36(6):503-16. doi: 10.1111/j.1600-0528.2008.00427.x. Epub 2008 Apr 14. PMID 18422711
- See also: Click here for more information about this study: A 2-year Community Trial of Fluoride Varnish for the Prevention of Early Childhood Caries in Aboriginal Children — http://www.caphd-acsdp.org/PDF/Aboriginal%20Preschool.pdf
- See also: Results of A Fluoride Varnish Trial to Prevent and Reduce Caries in Aboriginal Children — http://www.ncbi.nlm.nih.gov/pubmed/18422711?ordinalpos=9&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum